CLINICAL TRIAL: NCT04959786
Title: Effect of a Combination of Nitazoxanide, Ribavirin and Ivermectin Plus Zinc Supplement on the Clearance of COVID-19: Extension Study
Brief Title: MANS-NRIZ Trial for COVID-19 Treatment : Extension Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hatem Elalfy, professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mu-med-2020-26
Record Dates: First submitted 2021-07-01; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Ivermectin; Zinc

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION ARM (Experimental)
  Interventions: Drug: Ivermectin,ribavirin ,nitazoxanide and zinc
- standard of care (No Intervention)

INTERVENTIONS:
Drug: Ivermectin,ribavirin ,nitazoxanide and zinc — oral intake of the 3 drugs ivermectin ,ribavirin and nitazoxanide plus zinc
  Arms: INTERVENTION ARM

SUMMARY:
This search will focus on patients with COVID 19 infection this study is a prospective cohort study based on the analysis of response in comparative panel between two arm Nitazoxanide, Ribavirin and Ivermectin plus Zinc arm and other arm without any intervention as regards the safety and efficacy and cost effective result. Two years duration of the project would be enough to cover the stages of the work as shown below in the time plan. Initial stage of collecting materials and patients' clinical data, each patient will undergoes strict follow up period to reveal the clinical, laboratory and radiological response. The procedures are to be approved by the institutional ethical committee.

DETAILED DESCRIPTION:
This search will focus on patients with COVID 19 infection this study is a prospective cohort study based on the analysis of response in comparative panel between two arm Nitazoxanide, Ribavirin and Ivermectin plus Zinc arm and other arm without any intervention as regards the safety and efficacy and cost effective result. Two years duration of the project would be enough to cover the stages of the work as shown below in the time plan. Initial stage of collecting materials and patients' clinical data, each patient will undergoes strict follow up period to reveal the clinical, laboratory and radiological response. The procedures are to be approved by the institutional ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years

  * Laboratory-confirmed SARS-CoV- 2 infection
  * Hospitalized patients
* need reservoir mask for oxygen support
* need HFNC for oxygen support

Exclusion Criteria:

* Mechanical ventilations for oxygen support
* Inability to take oral medications
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Stabilization of oxygen | 28 days
  at room air more than 90%
In-hospital and 28-day mortality | 28 day

SECONDARY OUTCOMES:
Negative conversion of SARS-CoV- 2 by Day 28 | 28 day
Time to clinical improvement | 28 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Select A State Or Province, Egypt